CLINICAL TRIAL: NCT06908291
Title: A Cohort Study on the Development of a Standardized Scoring System for Breast Nodule Differential Diagnosis, Molecular Classification, and Neoadjuvant Chemotherapy Evaluation Using Photoacoustic/Ultrasound Imaging
Brief Title: Photoacoustic/Ultrasound Imaging for Breast Nodule Diagnosis, Molecular Classification, and Neoadjuvant Chemotherapy Response Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PA/US Breast Tumor
Record Dates: First submitted 2025-01-12; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: Breast Masses; Breast Cancer; Breast Cancer Treated with Neoadjuvant Chemotherapy
Keywords: Breast cancer; neoadjuvant chemotherapy; photoacoustic imaging; multi-modality imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breast nodules diagnosis cohort based on PA/US imaging (Experimental): Build a photoacoustic (PA) imaging (PAI) standardized scoring system to identify benign and malignant tumors, and use PAI to further determine the molecular classification of malignant breast tumors
  Interventions: Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system
- Participants with breast cancer planning to undergo NAC based on PA/US imaging (Experimental): Patients over 18 years of age with histopathologically confirmed breast cancer with clinical stage T2 or above (≥20 mm in diameter) and/or lymph node positivity and plan to undergo neoadjuvant chemotherapy.
  Interventions: Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system

INTERVENTIONS:
Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system — The multi-modal PA/US imaging system is equipped with a handheld PA/US probe, and able to provide data of dual-wavelength PA imaging of breat tomor and Ipsilateral axillary lymph nodes, in addition to real-time 2D PA/US imaging.

SUMMARY:
Photoacoustic (PA) imaging (PAI) emergerd as a rapidly evolving biomedical imaging modality, which combines the merits of optical imaging and ultrasound (US) imaging, and has a capacity in morphological, functional and molecular imaging, showing potential in visualizing superficial organs. The goal of this clinical trial is to build a PAI standardized scoring system to identify benign and malignant tumors, and use PAI to further determine the molecular classification of malignant breast tumors, and monitor the efficacy of neoadjuvant chemotherapy (NAC) in breast cancer. The main questions it aims to answer are:

1. How to build a standardized PA/US scoring system in differential diagnosis of benign and malignant tumors?
2. Can PAI precisely determine the molecular classification of breast tumors?
3. Can PAI systems predict the efficacy of NAC in breast cancer?

Participants will receive regular PA/US imaging examinations during four stages of NAC (before NAC, 2 Cycles, 4 Cycles and 6 Cycles). And the effectiveness of PA/US in predicting NAC for breast cancer at different time points will be evaluated.

DETAILED DESCRIPTION:
The multi-modality PA/US imaging system was built on a high-end commercial US platform and allowed real-time imaging of grey-scale US imaging, Color-Doppler US (CDUS) imaging and dual-wavelength PAI. The PA/US images were acquired using a hand-held probe integrated optical devices and US transducers. Researchers plan to recruit participants planning to undergo breast nodular surgery from the outpatient department of breast surgery in Peking Union Medical College Hospital. The patients are scheduled to receive multi-modality imaging examinations using the novel imaging system. First, conventional US scanning of the breast, including grey-scale US and CDUS, will be carried out by an experienced US operator. Afterwards, PA/US imaging will be implemented for breasts by the same operator. And the conventional ultrasound and photoacoustic information of the tumor will be assessed, including the tumor size, shape, boundary, calcificaition condition, the tumor blood flow and blood oxygenation. This clinical trial aims to address three key objectives: the development of a standardized PAI scoring system for distinguishing benign from malignant tumors, the application of PAI to assess the molecular classification of malignant breast tumors, and the use of PAI to monitor the efficacy of neoadjuvant chemotherapy (NAC) in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were above 18 years-old;
2. The patients were presented with a breast tumor, which were clearly shown on routine ultrasound; Biopsy or surgery of breast lesions was performed within 1 week and pathological diagnosis was obtained.
3. Patients agreed to participate in this experiment and signed the Subject Informed Consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Breast inflammation or local external injury;
3. The breast mass has been excised for biopsy.
4. Poor photoacoustic imaging effect.
5. Deep lesion location (>3.5 cm)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Establish Photoacoustic/Ultrasound Standardized Scoring System for Differentiating Benign and Malignant Breast Masses | From enrollment to the end of treatment at 2 year
  In this study, 300 patients who planned to undergo breast nodule surgery were enrolled. Tumor size, shape, boundary, calcification condition, peripheral vascular morphology, blood oxygen saturation (SO2), internal blood flow richness, blood oxygen semi-quantitative score will be measured in the standardized scoring system, and these photoacoustic and ultrasound parameters will be used to classify the mass as benign or malignant.
Predict the Precise Molecular Subtypes of Malignant Breast Masses Using Photoacoustic/Ultrasound Parameters | From enrollment to the end of treatment at 2 years
  In this study, the same cohort as the first one will be used. Tumor size, shape, boundary, calcification condition, peripheral vascular morphology, blood oxygen saturation (SO2), internal blood flow richness, blood oxygen semi-quantitative score will be measured, and these photoacoustic and ultrasound parameters will be used to predict the precise molecular subtypes of malignant breast masses.
Evaluate Tumor Residual and Lymph Node Burden in Breast Cancer after Neoadjuvant Therapy | From enrollment to the end of treatment at 3 years
  This study included 250 breast cancer patients confirmed by needle bioposy, with clinical stage T2 or above (diameter ≥20 mm) and/or with positive lymph nodes, who were to undergo neoadjuvant chemotherapy. Tumor size, shape, boundary, calcification condition, vascular richness, vascular morphology, blood oxygen saturation will be measured as indicators to predict pathological complete response (pCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided